CLINICAL TRIAL: NCT07037732
Title: Circulating B-cell, Drug and Anti-drug Antibodies Monitoring in Patients Treated With Rituximab for Autoimmune Disorders : the MONIRITUX Study
Brief Title: Circulating B-cell, Drug and Anti-drug Antibodies Monitoring in Patients Treated With Rituximab for Autoimmune Disorders
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Immuno01
Record Dates: First submitted 2025-05-23; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Cytopenia; Connective Tissue Disorder; Systemic Vasculitis
MeSH Terms: conditions — Connective Tissue Diseases; Systemic Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Autoimmune cytopenia (immune thrombocytopenia or hemolytic anemia): Blood CD19+, CD27+, and CD38+ B-cell reconstitution, circulanting rituximab level or the presence of circulating anti-rituximab antibodies will be compared in patients experiencing clinical relapse and those who will remain stable over time.
- Connective tissu disorder (SLE, myopathie, RA…): Blood CD19+, CD27+, and CD38+ B-cell reconstitution, circulanting rituximab level or the presence of circulating anti-rituximab antibodies will be compared in patients experiencing clinical relapse and those who will remain stable over time.
- Systemic vasculitis (ANCA, essential cryoglobulinemia): Blood CD19+, CD27+, and CD38+ B-cell reconstitution, circulanting rituximab level or the presence of circulating anti-rituximab antibodies will be compared in patients experiencing clinical relapse and those who will remain stable over time.

SUMMARY:
The MONIRITUX study aimed to evaluate whether monitoring (i) circulating B-cell reconstitution or (ii) serum rituximab levels could help identify relapse of autoimmune diseases in patients treated with rituximab. Retrospective data suggest that B-cell reconstitution or the appearance of anti-drug antibodies are associated with rituximab's failure to prevent relapses (i.e. rheumatoid arthritis, systemic lupus erythematosus, autoimmune cytopenia...). According to the routine care provided by our institution, patients undergoing rituximab therapy are monitored every three months during the first year after treatment induction and every six months thereafter. At each clinical visit, a blood test is performed to quantify total gammaglobulins, IgG and CD19+ cells (along with other tests depending on the disease). This study will use the remaining blood in the tubes from routine care to quantify CD27+ and CD38+ B cells, as well as serum rituximab and anti-rituximab antibodies, during the first year of follow-up. The primary outcome will be to identify risk factors for clinical relapse according to circulating B-cell or rituximab status.

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergo rituximab treatment according to routine care and having one of the following disorder:
* primary immune thrombocytopenia
* primary autoimmune hemolytic anemia
* systmic lupus erythematous
* systemic sclerosis
* rheumatoid arthritis
* inflammatory myopathy
* ANCA associated vasculitis
* Cryoglobulinemic vasculitis

Exclusion Criteria:

* Patients undergoing multiple immunosuppressive drugs because of refractory disease or concomitant hemopathy or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who undergo rituximab treatment according to routine care and having one of the following disorder:
  * primary immune thrombocytopenia
  * primary autoimmune hemolytic anemia
  * systmic lupus erythematous
  * systemic sclerosis
  * rheumatoid arthritis
  * inflammatory myopathy
  * ANCA associated vasculitis
  * Cryoglobulinemic vasculitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Patients with (Immune Thrombocytopenia) ITP | At each consultation during 5 years
  Hematologic relapse described as a drop in platelet count below 20 G/L following a remission phase of at least 3 months with platelet count greater than 50 G/L.
Patients with AIHA Autoimmune Hemolytic Anemia. | At each consultation during 5 years
  Hematologic relapse described as a drop in hemoglobin level below 10 g/dL (with a lost of at least 2 g/dL from baseline) in association with hemolysis after e remission of at least 3 months
Patients with inflammatory myopathy | At each consultation during 5 years
  Clinical relase defined as a confirmed muscular (myalgia associated with at least one from the following : increase CK levels, new or worsening electromyography, new or worsening muscle inflammation on MRI), joint or pulmonary new symptoms related to myositis
Patients with systemic lupus erythematous : | At each consultation during 5 years
  Clinical relapse defined as an increase by 4 points in the SLEDAI (systemic lupus erythematous disease activity index) score
Patients with systemic vasculitis | At each consultation during 5 years
  Clinical relapse defined as an increase by 1 points in the Birmingham vasculitis (BVAS) score

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, Alpes Maritimes, France